CLINICAL TRIAL: NCT02470247
Title: IPC-Angio Trial : Interest of Remote Ischemic Preconditioning for Prevention of Contrast Medium-induced Nephropathy (Post-diagnostic Imaging) in Patients at High Risk of Contrast-induced Nephropathy
Brief Title: Interest of Remote Ischemic Preconditioning for Prevention of Contrast Medium-induced Nephropathy in High Risk Patients
Acronym: IPC-Angio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 35RC14_9899_IPC-Angio Trial; 150058B-11 (Other: ANSM); 15/07-969 (Other: Comité de Protection des Personnes); 2015-A00076-43 (Other: ANSM)
Record Dates: First submitted 2015-06-05; First posted 2015-06-12 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Nephropathy
Keywords: Transcatheter Aortic Valve Implantation
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remote ischemic preconditioning (Experimental): Remote Ischemic Preconditioning (RIPC) is accomplished by performing 4 cycles of alternating 5-minute inflation and 5-minute deflation of a standard upper-arm blood pressure cuff, to induce transient and repetitive arm ischemia and reperfusion.
  RIPC will be started just before the CTA, and the time between the last inflation cycle and the beginning of the CTA will be less than 45 minutes.
  Interventions: Other: Remote Ischemic Preconditioning (RIPC)
- SHAM remote ischemic preconditioning (Sham Comparator): The SHAM Remote Ischemic Preconditioning ("SHAM" RIPC) will be carried out with the same number of cycles that the RIPC but cuff will be inflated to the diastolic pressure of the subject and the cuff will be deflated to10 mmHg in order to maintain a non- ischemic compression (blind patient protocol).
  Interventions: Other: SHAM Remote Ischemic Preconditioning (SHAM RIPC)

INTERVENTIONS:
Other: Remote Ischemic Preconditioning (RIPC) — RIPC is accomplished by performing 4 cycles of alternating 5-minute inflation and 5-minute deflation of a standard upper-arm blood pressure cuff, to induce transient and repetitive arm ischemia and reperfusion.
  RIPC will be started just before the CTA, and the time between the last inflation cycle and the beginning of the CTA will be less than 45 minutes.
  Arms: Remote ischemic preconditioning
Other: SHAM Remote Ischemic Preconditioning (SHAM RIPC) — The SHAM Remote Ischemic Preconditioning ("SHAM" RIPC) will be carried out with the same number of cycles that the RIPC but cuff will be inflated to the diastolic pressure of the subject and the cuff will be deflated to10 mmHg in order to maintain a non- ischemic compression (blind patient protocol).
  Arms: SHAM remote ischemic preconditioning

SUMMARY:
Diagnostic imaging for vascular investigations and endovascular procedures frequently require the use of contrast medium. Besides contrast medium-induced hypersensitivity, an acute kidney injury can appear: the contrast-induced nephropathy (NPCI).

NPCI is associated with an increase of patients' morbidity and mortality. One of the conventional methods proposed to limit this NPCI is an oral administration of N-acetylcysteine (NAC) associated with hydration performed 12 hours before and 12 hours after the injection. However, in some patients this method cannot be performed due to a high risk of heart failure although they are generally at high risk of NPCI.

Recently, it has been shown, in a randomized trial, that remote ischemic preconditioning (several cycles of upper-arm ischemia-reperfusion with a pressure cuff inflator) associated with hydratation and NAC reduced the occurrence of NPCI after a coronary angiography as compared with NAC and hydration only. .

We hypothesized that the use of RIPC in patients at high risk of NPCI and who cannot receive NAC and hydratation (e.g. patients with aortic stenosis and eligible for Transcatheter Aortic Valve Implantation (TAVI)) could be promising.

DETAILED DESCRIPTION:
Study design :

Prospective, single-center, randomized, controlled, single-blind, with RIPC procedure (Pre-CI) versus "SHAM" ischemic preconditioning (SHAM Pre -CI) (control). This test will follow the CONSORT Statement (http://www.consort-statement.org/).

This is a randomized, controlled, single-blind trial, assessing the incidence of NPCI (after a CTA ) between two group of patients, one receiving RIPC procedure and the other group receiving a "SHAM" RIPC (control group).

RIPC is accomplished by performing 4 cycles of alternating 5-minute inflation and 5-minute deflation of a standard upper-arm blood pressure cuff, to induce transient and repetitive arm ischemia and reperfusion.

RIPC will be started just before the CTA, and the time between the last inflation cycle and the beginning of the CTA will be less than 45 minutes. The "SHAM" RIPC will be carried out with the same number of cycles that the RIPC but cuff will be inflated to the diastolic pressure of the subject and the cuff will be deflated to10 mmHg in order to maintain a non- ischemic compression (blind patient protocol).

Main objective :

To assess the efficacy of remote ischemic preconditioning (RIPC) in preventing contrast-induced nephropathy (NPCI) after injected CT scanner in patients at high risk of NPCI.

Secondary objectives :

1. To assess the effects of RIPC on a second marker of renal failure (Cystatin C ) ;
2. To determine the pathophysiological mechanisms involved in the RIPC (role of oxidative stress ; for the first 40 patients) ;
3. To assess the effect of RIPC on renal function after a second injection of contrast-medium during coronary angiography performed 2 to 4 days after the injected CTA ;
4. To assess the tolerance of RIPC procedure ;
5. To assess the impact on mortality at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years, no upper age limit ;
* Patient which may hospitalized for a medical check-up before a percutaneous aortic valve implantation (CTA and coronarography);
* Patient at risk for NPCI defined by a Mehran risk classification system ≥11 (Annexe 2) ;
* Willing to provide free and informed written consent

Exclusion Criteria:

* Pathology of the upper-limbs limiting the use of the cuff (bilateral amputation, arteriovenous fistula);
* Critical renal disease requiring hemodialysis ;
* Person who is not affiliated to a health care system insurance
* Inability to understand the instructions of the study;
* Absolute contraindication to of iodinated contrast medium injection (anaphylactic shock history to contrast media, especially Xenetix, clearance (MDRD) less than 30mL/min/1.73m2) ;
* Pregnancy
* Simultaneous participation in other protocol;
* Person with legal protection, person deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-10-06 (Actual); Primary Completion 2017-08-24 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of NPCI | 48 hours
  Incidence of NPCI defined as an increase in serum creatinine ≥ 0.5 mg / dL or a relative increase of 25 % above baseline at 48 hours after contrast medium exposure.

SECONDARY OUTCOMES:
Cystatin C | 2 days
  Changes of serum Cystatin C between day 0 and day 1, and day 0 and day 2.
Oxydative stress | 24 hours
  Changes in markers of oxydative stress (in the first 40 patients included) :
  * at day 0, after the RIPC procedure or SHAM-RIPC procedure (+ 5 min) before CTA ;
  * after CTA (+ 30 min) and 24 hours after CTA (day 1).
Renal function | 6 days
  Changes in serum creatinine and Cystatin C between day 0 and measured values after coronarography (day 6 ).
Pain | Day 0
  A standardized pain scale (ranged from 0 to 10; 0 : no pain; 10 : maximum of pain).
Mortality | 6 months
  Assessment of mortality at six months.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Mahe, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, Britanny, France

REFERENCES:
- [Result] Belabbas D, Koch C, Chaudru S, Lederlin M, Laviolle B, Le Pabic E, Boulmier D, Heautot JF, Mahe G. Effects of Remote Ischemic Pre-Conditioning to Prevent Contrast-Induced Nephropathy after Intravenous Contrast Medium Injection: A Randomized Controlled Trial. Korean J Radiol. 2020 Nov;21(11):1230-1238. doi: 10.3348/kjr.2019.0916. Epub 2020 Jul 27. PMID 32729273
- [Result] Koch C, Chaudru S, Lederlin M, Jaquinandi V, Kaladji A, Mahe G. Remote Ischemic Preconditioning and Contrast-Induced Nephropathy: A Systematic Review. Ann Vasc Surg. 2016 Apr;32:176-87. doi: 10.1016/j.avsg.2015.10.017. Epub 2016 Jan 21. PMID 26802296